CLINICAL TRIAL: NCT04178265
Title: Electroacupuncture Improves Pain and Wrist Functionality in Patients Undergoing Rehabilitation Therapy After Arthroscopic Repair for Triangular Fibrocartilage Complex (TFCC) Tears.
Brief Title: Electroacupuncture Improves Pain and Wrist Functionality
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMUH108-REC2-057
Record Dates: First submitted 2019-11-07; First posted 2019-11-26 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Electroacupuncture
Keywords: electroacupuncture; triangular fibrocartilage complex tears; TFCC tears; pain; wrist functionality
MeSH Terms: conditions — Pain | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electroacupuncture group (Experimental): At the 4th week after surgery, electroacupuncture was performed, and the activity of wrist joint on the affected side was performed at same time, and at a frequency of three times per week for four weeks, for a total of twelve times.
  Acupoint selection: needles were inserted to Kunlun(BL60), Yanglingquan (GB34), Sanyinjiao(SP6), Taixi (KI 3) contralateral to the operated leg and deqi sensation elicited at acupoints.
  Interventions: Other: Electroacupuncture
- Control group (No Intervention): At the 4th week after surgery, only the activity of wrist joint on the affected side was performed, and at a frequency of three times per week for four weeks, for a total of twelve times.

INTERVENTIONS:
Other: Electroacupuncture — needles were inserted to Kunlun(BL60), Yanglingquan (GB34), Sanyinjiao(SP6), Taixi (KI 3) contralateral to the operated leg and deqi sensation elicited at acupoints.
  Arms: Electroacupuncture group

SUMMARY:
Triangular Fibrocartilage Complex (TFCC) is the main stable structure of the distal ulnar joint (DRUJ), and the damage of the triangular fibrocartilage complex is the most common cause of pain in the ulnar side of the wrist in the young athlete population. Once TFCC is injured, arthroscopic surgery is a common repair method. And, the postoperative goal is to restore the function of the forearm and the mobility of the wrist joint. Therefore, rehabilitation treatment is the key. However, postoperative patients often delay rehabilitation therapy due to pain, resulting in stiffer wrist joints. In recent years, electroacupuncture(EA) has been widely used to relieve pain after surgery, and many studies have confirmed that it is effective. And it is already an alternative to postoperative pain relief. The investigators hope that by electroacupuncture, the investigators can help patients reduce pain, increase joint mobility, and make patients willing to start rehabilitation therapy, reduce joint stiffness, and restore wrist function as soon as possible, which will help patients return to work and normal life early.

DETAILED DESCRIPTION:
Methods:

It is expected that 30 patients will be randomly assigned to the following groups: electroacupuncture group, control group without EA. Two groups of subjects started to rehabilitation therapy at a hospital or clinic at the 4th week after surgery.

Mode of operation:

Electroacupuncture group: At the 4th week after surgery, electroacupuncture was performed, and the activity of wrist joint on the affected side was performed at same time, and at a frequency of three times per week for four weeks, for a total of twelve times.

Control group: At the 4th week after surgery, only the activity of wrist joint on the affected side was performed, and at a frequency of three times per week for four weeks, for a total of twelve times.

Acupoint selection: needles were inserted to Kunlun(BL60), Yanglingquan (GB34), Sanyinjiao(SP6), Taixi (KI 3) contralateral to the operated leg and deqi sensation elicited at acupoints.

Data collection:

The evaluator does not know the patient group to achieve a single blind effect.

1. Use the visual analog scale (VAS) to assess the patient's pain level
2. Use the Disabilities of the Arm, Shoulder and Hand(DASH) to assess the patient's pain and the inability.
3. The degrees of wrist mobility were measured.
4. Three time points were recorded: before the first electroacupuncture (4th week after surgery, when removing fixation), after the 6th, 12th (last) electroacupuncture.
5. Record the time point of the wrist joint recovery function and return to the workplace.

ELIGIBILITY:
Inclusion Criteria:

1. Orthopedic specialist diagnoses tearing of the triangular fibrocartilage complex and undergoes arthroscopic surgery
2. Age between 19 and 60 years old

Exclusion Criteria:

1. serious heart rhythm
2. epilepsy
3. Severe pulmonary heart disease
4. History of mental illness
5. received acupuncture treatment 1 month ago

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-05-06 (Actual); Primary Completion 2020-05-05 (Estimated); Study Completion 2020-05-05 (Estimated)

PRIMARY OUTCOMES:
Range of wrist motion | 4 weeks
  The degrees of wrist mobility measured with a goniometer, including flexion, extension, supination, pronation, ulnar deviation, radial deviation, and higher degrees mean a better outcome.

SECONDARY OUTCOMES:
Disabilities of the Arm, Shoulder and Hand(DASH) | 4 weeks
  Assess the patient's pain and the inability, the DASH consists mainly of a 30-item disability/symptom scale, scored 0 (no disability) to 100.

CONTACTS AND LOCATIONS:
Overall Officials: Yung-Cheng Chiu, MD, Study Director — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, No. 2, Yude Rd, North District, Taichung City, Taiwan

IPD SHARING:
Plan to Share IPD: No